CLINICAL TRIAL: NCT05153577
Title: Fresh Start: Increasing Produce Access and Intake Among WIC-eligible Children in West Philadelphia
Brief Title: Fresh Start: Increasing Early Produce Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-018757
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Food Insecurity
Keywords: WIC

STUDY DESIGN:
Intervention Model Description: Potential subjects will initially be recruited from a list of 30 parents who participated in the previous IRB-exempt, qualitative study (IRB 20-017497 - Fresh Start) and consented to be re-contacted for future studies. The remaining subjects will be recruited from a list of families who received a WIC prescription for their child(ren) from a provider at the Children's Hospital of Philadelphia (CHOP) Cobbs Creek between 2019-2020; this list was obtained via IT query of Epic for our prior study. No medical records will be accessed for screening for this study. Potential subjects will be screened using the protocol inclusion and exclusion criteria during the initial recruitment call.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Free produce box (Active Comparator): Participants receive free weekly produce boxes for the first 4 weeks of the study and are then randomized to pay $5 per box (with continued free weekly delivery) for the remaining 4 weeks of the study.
  Interventions: Other: Group A: $5 produce box
- Group B: Free produce box (Active Comparator): Participants receive free weekly produce boxes for the first 4 weeks of the study and are then randomized to pay $10 per box (with continued free weekly delivery) for the remaining 4 weeks of the study.
  Interventions: Other: Group B: $10 produce box

INTERVENTIONS:
Other: Group A: $5 produce box — Participants receive free weekly produce boxes delivered to their home for the first 4 weeks of the study and are then randomized to pay $5 per box (with continued free weekly delivery) for the remaining 4 weeks of the study. Participants also complete survey at the beginning, middle, and end of the produce delivery program.
  Arms: Group A: Free produce box
Other: Group B: $10 produce box — Participants receive free weekly produce boxes delivered to their home for the first 4 weeks of the study and are then randomized to pay $10 per box (with continued free weekly delivery) for the remaining 4 weeks of the study. Participants also complete survey at the beginning, middle, and end of the produce delivery program.
  Arms: Group B: Free produce box

SUMMARY:
Nearly 22% of children in Philadelphia live in food-insecure (FI) households, often leading to reliance on inexpensive, nutrient-poor foods and associated poor health outcomes. Despite this, utilization of food benefit programs is often low, including the Special Supplemental Nutrition Program Women, Infants, and Children (WIC) Farmer's Market Nutrition Program (FMNP). In the prior qualitative study, Investigators found that parents desire to increase their children's intake of produce but face many barriers to produce access; caregivers described a preference for delivery-based, low-or-no cost food programs to increase produce access and intake among children. This pilot trial seeks to assess the effectiveness of a short-term, tiered-fee produce delivery program in retaining participants and increasing produce access and intake among families with WIC-eligible children

DETAILED DESCRIPTION:
Investigators are piloting a produce box delivery program to approximately 50 WIC-eligible, low-income families in West Philadelphia in partnership with the Farm to Families Initiative (St. Christopher's Foundation for Children) and Food Connect, a local food delivery program. Both partnerships have been previously established and are maintained through the Office of Community Relations. The program will be 8 weeks in duration; in the first 4 weeks, all families will receive a free, weekly produce box from Farm to Families. In the second two weeks, the 50 families will be randomized into two groups, each with 25 participants. One group will be asked to pay $5 for the produce box and the other group will pay $10, using food benefits or their own income. Recipes that include foods in the produce box will be included with the delivery along with children's activities (books, coloring pages, card games, etc.) related to fruits and vegetables. Participating parents will complete three online surveys throughout the program. These pre-, mid-, and post-intervention surveys will assess the effect of the program and participant satisfaction.

The expected goals are to:

1. Evaluate the effect of different pricing models on participation of low-income, WIC-eligible families in a produce delivery program
2. Evaluate the efficacy of a low-cost produce delivery program to increase perceived intake of produce among low-income young children.
3. Evaluate efficacy of a low-cost produce delivery program to increase perceived access to produce among low-income families in West Philadelphia.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

1. Be over 18 years of age
2. Be the parent or guardian for children ages 0 to 5 years of age who receive or are eligible to receive WIC benefits
3. Be the parent or guardian for children ages 0 to 5 years of age who receive pediatric care at CHOP Primary Care - Cobbs Creek
4. Live or have access to an address where packages can be delivered
5. Have access to an electronic device and internet in order to access the online produce box ordering portal
6. Be willing to complete three 10-15 minute surveys throughout the intervention either online or via telephone
7. Consent to have their contact information shared with Farm to Families and Food Connect

Exclusion Criteria:

Subjects must not:

1. Be participating in another intervention which provides produce just prior to or simultaneous with participation in this study (e.g. Farm Food Box Program, etc.)
2. Be subjects who, in the opinion of the Investigator(s), may be non-compliant with study schedules or procedures Subjects that do not meet all of the enrollment criteria may not be enrolled. Any violations of these criteria must be reported in accordance with IRB Policies and Procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Number of participants in both groups who continue to participate in the program weekly in different pricing models | 8 weeks
  Participant ordering in each group will be tracked weekly in RedCap for week 1, 2, 3, 4, 5, 6, 7, and 8.

SECONDARY OUTCOMES:
Evaluate the impact of the produce delivery program on perceived intake and enjoyment of fruits and vegetables | Up to 6 months
  The impact of the produce delivery program on perceived intake and enjoyment of fruits and vegetables will be measured using open-ended questions and 5-point Likert scale pre-enrollment, at midpoint during weeks 4-6, and at the end of the intervention after week 8. The measures of the scale include (1)Never, (2)Rarely, (3)Sometimes, (4)Often, and (5) Always.
Assess the efficacy of the produce delivery program in improving perceived diet | Up to 6 months
  The efficacy of the produce delivery program in improving perceived diet of participants and their children will be measured using open-ended questions and 5-point Likert scale pre-enrollment, at midpoint during weeks 4-6, and at the end of the intervention after week 8. The measures of the scale include (1) Strongly Disagree, (2) Disagree, (3) Neither Agree or Disagree, (4) Agree, and (5) Strongly Agree.
Evaluate the efficacy of the produce delivery program in improving perceived produce access, including attainability and cost, among the study population | Up to 6 months
  The efficacy of the produce delivery program in improving perceived produce access will be measured using open-ended questions and 5-point Likert scale pre-enrollment, at midpoint during weeks 4-6, and at the end of the intervention after week 8. The measures of the scale include (1) Strongly Disagree, (2) Disagree, (3) Neither Agree or Disagree, (4) Agree, and (5) Strongly Agree.
Assess self-efficacy among the study population in regards to preparing home-cooked meals, particularly with fruits and vegetables. | Up to 6 months
  Self-efficacy among the study population in regards to preparing home-cooked meals, particularly with fruits and vegetables will be measured using open-ended questions and 5-point Likert scale pre-enrollment, at midpoint during weeks 4-6, and at the end of the intervention after week 8. The measures of the scale include (1) Strongly Disagree, (2) Disagree, (3) Neither Agree or Disagree, (4) Agree, and (5) Strongly Agree.
Evaluate for changes in reported food insecurity among the stated study population. | Up to 6 months
  Investigators will evaluate for food insecurity using a validated food insecurity screening tool pre-enrollment, at midpoint during weeks 4-6, and at the end of the intervention after week 8. Questions in the tool include (1)In the past 30 days, we worried that our food would run out before we got money to buy more; (2) In the past 30 days, the food we bought ran out and we didn't have money to get more; and (3) In the past 30 days, we couldn't afford to eat balanced meals. Response options include (1) Often True, (2) Sometimes True, and (3) Never True.
Determine if the Fresh Start produce delivery program leads to changes in food purchasing patterns among the study population. | Up to 6 months
  Impact of the produce delivery program leading to changes in food purchasing patterns will be measured using open-ended questions and 4-point Likert scale at midpoint during weeks 4-6 and at the end of the intervention after week 8. The measures of the scale include (1) I Buy Less, (2) I Buy The Same Amount, (3) I Buy More, and (4) Does Not Apply/I Have Never Bought This.
Assess participant satisfaction with the Fresh Start produce delivery program | Up to 6 months
  Investigators will assess participant satisfaction with the Fresh Start produce delivery program will be measured using open-ended questions and 5-point Likert scale at midpoint during weeks 4-6 and at the end of the intervention after week 8. The measures of the scale include (1)Very Unhappy, (2) Unhappy, (3)Neutral, (4)Happy, and (5) Very Happy.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Cullen, MD, MPH, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
N/A - The IPD will only be utilized by the researchers currently on the project.

REFERENCES:
- [Background] Kim SA, Moore LV, Galuska D, Wright AP, Harris D, Grummer-Strawn LM, Merlo CL, Nihiser AJ, Rhodes DG; Division of Nutrition, Physical Activity, and Obesity, National Center for Chronic Disease Prevention and Health Promotion, CDC. Vital signs: fruit and vegetable intake among children - United States, 2003-2010. MMWR Morb Mortal Wkly Rep. 2014 Aug 8;63(31):671-6. PMID 25102415
- [Background] Di Noia J, Byrd-Bredbenner C. Determinants of fruit and vegetable intake in low-income children and adolescents. Nutr Rev. 2014 Sep;72(9):575-90. doi: 10.1111/nure.12126. Epub 2014 Aug 4. PMID 25091630
- [Background] Krolner R, Rasmussen M, Brug J, Klepp KI, Wind M, Due P. Determinants of fruit and vegetable consumption among children and adolescents: a review of the literature. Part II: qualitative studies. Int J Behav Nutr Phys Act. 2011 Oct 14;8:112. doi: 10.1186/1479-5868-8-112. PMID 21999291
- [Background] COUNCIL ON COMMUNITY PEDIATRICS; COMMITTEE ON NUTRITION. Promoting Food Security for All Children. Pediatrics. 2015 Nov;136(5):e1431-8. doi: 10.1542/peds.2015-3301. PMID 26498462
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Food and Nutrition Board; Committee to Review WIC Food Packages. Review of WIC Food Packages: Improving Balance and Choice: Final Report. Washington (DC): National Academies Press (US); 2017 May 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK435902/ PMID 28605175
- [Background] Anderson JV, Bybee DI, Brown RM, McLean DF, Garcia EM, Breer ML, Schillo BA. 5 a day fruit and vegetable intervention improves consumption in a low income population. J Am Diet Assoc. 2001 Feb;101(2):195-202. doi: 10.1016/S0002-8223(01)00052-9. PMID 11271692
- [Background] Kropf ML, Holben DH, Holcomb JP Jr, Anderson H. Food security status and produce intake and behaviors of Special Supplemental Nutrition Program for Women, Infants, and Children and Farmers' Market Nutrition Program participants. J Am Diet Assoc. 2007 Nov;107(11):1903-8. doi: 10.1016/j.jada.2007.08.014. PMID 17964309
- [Background] Di Noia J, Monica D, Sikorskii A, Nelson J. Pilot Study of a Farm-to-Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) Intervention Promoting Vegetable Consumption. J Acad Nutr Diet. 2021 Oct;121(10):2035-2045. doi: 10.1016/j.jand.2020.12.020. Epub 2021 Jan 22. PMID 33487590
- [Background] Lagisetty P, Flamm L, Rak S, Landgraf J, Heisler M, Forman J. A multi-stakeholder evaluation of the Baltimore City virtual supermarket program. BMC Public Health. 2017 Oct 23;17(1):837. doi: 10.1186/s12889-017-4864-9. PMID 29061141
- [Background] Townsend MS, Kaiser LL, Allen LH, Joy AB, Murphy SP. Selecting items for a food behavior checklist for a limited-resource audience. J Nutr Educ Behav. 2003 Mar-Apr;35(2):69-77. doi: 10.1016/s1499-4046(06)60043-2. PMID 12725713
- [Background] Couch SC, Glanz K, Zhou C, Sallis JF, Saelens BE. Home food environment in relation to children's diet quality and weight status. J Acad Nutr Diet. 2014 Oct;114(10):1569-1579.e1. doi: 10.1016/j.jand.2014.05.015. Epub 2014 Jul 23. PMID 25066057
- [Background] Lahne J, Wolfson JA, Trubek A. Development of the Cooking and Food Provisioning Action Scale (CAFPAS): A new measurement tool for individual cooking practice. Food Qual Prefer. 2017;62(July):96-105. doi:10.1016/j.foodqual.2017.06.022
- [Background] Hager ER, Quigg AM, Black MM, Coleman SM, Heeren T, Rose-Jacobs R, Cook JT, Ettinger de Cuba SA, Casey PH, Chilton M, Cutts DB, Meyers AF, Frank DA. Development and validity of a 2-item screen to identify families at risk for food insecurity. Pediatrics. 2010 Jul;126(1):e26-32. doi: 10.1542/peds.2009-3146. PMID 20595453
- [Derived] Joshi P, Van Remortel BJ, Rameswaran J, Cullen DL. Effect of Price on Women, Infants, and Children-Eligible Caregiver Participation in a Produce Program: A Randomized Trial. Acad Pediatr. 2025 Nov-Dec;25(8):102884. doi: 10.1016/j.acap.2025.102884. Epub 2025 Jul 9. PMID 40645578
- See also: National Cancer Institute. Usual Dietary Intakes: Food Intakes, U.S. Population, 2007-10. — https://epi.grants.cancer.gov/diet/usualintakes/national-data-usual-dietary-intakes-2007-to-2010.pdf
- See also: Coleman-Jensen A, Rabbitt MP, Gregory CA, Singh A. Household Food Security in the United States in 2019. — http://www.ers.usda.gov/publications/pub-details/?pubid=99281
- See also: Feeding America. Map the Meal Gap. Child Food Insecurity in Philadelphia County. Accessed February 20, 2021. — https://map.feedingamerica.org/county/2018/child/pennsylvania/county/philadelphia/
- See also: US Department of Agriculture, Food and Nutrition Service. WIC FMNP FY 2018 FNS-203 Report. — https://www.fns.usda.gov/fmnp/wic-farmers-market-nutrition-program